CLINICAL TRIAL: NCT01504815
Title: Phase III Randomized Study With Cisplatinum and Conventional or Adaptive High Dose Radiotherapy for Advanced Head and Neck Cancer
Brief Title: Adaptive Radiation Treatment for Head and Neck Cancer
Acronym: ARTFORCE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Karolinska Institutet (Other); Maastricht Radiation Oncology (Other); Institut Catala de Salut (Other Government); The Christie NHS Foundation Trust (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); UMC Utrecht (Other); European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M11ART
Record Dates: First submitted 2011-12-15; First posted 2012-01-05 (Estimated); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
Keywords: advanced head and neck cancer; adaptive radiotherapy; cisplatinum
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cisplatinum + conventional RT (Active Comparator): Cisplatinum 100mg/m2 on days 1, 22 and 43, with conventional RT 70 Gy in 7 weeks
  Interventions: Drug: cisplatinum; Radiation: Conventional radiotherapy
- Cisplatinum + adaptive high dose RT (Experimental): Cisplatinum, 100 mg/m2 on days 1, 22 and 43 with adaptive high dose RT to 84 Gy max on 50% uptake GTV in 7 weeks
  Interventions: Drug: cisplatinum; Radiation: Adaptive radiotherapy

INTERVENTIONS:
Drug: cisplatinum — i.v. 100 mg/m2 on days 1, 22 and 43 of radiotherapy
Radiation: Conventional radiotherapy — conventional radiotherapy, 70Gy in 7 weeks
  Arms: Cisplatinum + conventional RT
Radiation: Adaptive radiotherapy — adaptive high dose radiotherapy up to 84 Gy max on 50% uptake GTV in 7 weeks
  Arms: Cisplatinum + adaptive high dose RT

SUMMARY:
This Phase III trial aims to:

Explore the impact of pre-treatment information and radiation dose redistribution on locoregional control in patients with locally advanced SCCHN.

The dose to the primary tumor with margins, based upon PET and CT information, will be inhomogeneously increased to a tumor dose between 70 and 84 Gy with decreasing dose towards the edges of the irradiated area.

To determine the toxicity of combined modality treatment (cisplatin) with standard dose distribution versus combined modality treatment (cisplatin) with adaptive inhomogeneous radiation dose distribution.

ELIGIBILITY:
Inclusion Criteria:

* biopsy-confirmed squamous cell carcinoma of the oropharynx, oral cavity or hypopharynx
* stage III/IV, T3-4, Nx M0
* < 70 yrs
* glomerular filtration rate (GFR) >60
* WHO 0-1
* no previous malignancies except for adequately treated basal cell carcinoma of the skin and carcinoma in situ of the cervix
* adequate bone marrow function, adequate hepatic function,informed consent
* >18 years

Exclusion Criteria:

* expected failure from follow-up
* previous malignancies except for adequately treated basal cell carcinoma of the skin and carcinoma in situ of the cervix
* expected inability to complete either one of the treatment arms
* pregnancy or lactation
* patients (m/f) with reproductive potential not implementing adequate contraceptive measures
* prior surgery, radiotherapy or chemotherapy for this tumor
* contraindications or serious concomitant diseases preventing the safe administration of chemotherapy and/or radiotherapy or are likely to interfere with the study assessments
* known active symptomatic fungal, bacterial and/or viral infections including HIV
* concomitant (or with 4 weeks before randomisation) administration of any other experimental drug
* concurrent treatment with any other anti-cancer therapy
* prior treatment with one or more of the active compounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2012-09-07 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
locoregional recurrence-free survival | 2 years
number of patients with grade 3 toxicity or more | 2 years

SECONDARY OUTCOMES:
Quality of Life assessment | 2 years
swallowing preservation | 1 year
  Tube feeding dependency at one year
progression free survival | 2 years
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Olga Hamming-Vrieze, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (9):
- Gustave Roussy Cancer Institute, Villejuif, France
- Netherlands (5):
  - Netherlands Cancer Institute, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Maastro Clinic, Maastricht
  - Erasmus Medical Centre, Rotterdam
  - University Medical Centre Utrecht, Utrecht
- University Hospital Vall d'Hebron, Barcelona, Spain
- Karolinska Institute, Stockholm, Sweden
- Christie Hospital NHS Trust, Manchester, United Kingdom

REFERENCES:
- [Derived] Heukelom J, Hamming O, Bartelink H, Hoebers F, Giralt J, Herlestam T, Verheij M, van den Brekel M, Vogel W, Slevin N, Deutsch E, Sonke JJ, Lambin P, Rasch C. Adaptive and innovative Radiation Treatment FOR improving Cancer treatment outcomE (ARTFORCE); a randomized controlled phase II trial for individualized treatment of head and neck cancer. BMC Cancer. 2013 Feb 22;13:84. doi: 10.1186/1471-2407-13-84. PMID 23433435